CLINICAL TRIAL: NCT05073666
Title: Prevalence and Risk Factors of Chronic Thrombo-embolic Disease After a Pulmonary Embolism Event The PACTE Registry
Brief Title: Prevalence and Risk Factors of Chronic Thrombo-embolic Disease After a Pulmonary Embolism Event
Acronym: PACTE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Cardio02
Record Dates: First submitted 2021-09-08; First posted 2021-10-11 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Emboilism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pulmonary embolism: Patients with a recent pulmonary embolism event will be followed for 6 months and will benefit of routine tests (Lung scintigraphy, venous echo doppler, d- dimers measurement) in order to determine chronic thrombo-embolic disease prevalence and its risk factors.
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — NO INTERVENTION

SUMMARY:
Venous thromboembolic disease (VTE) is a common clinical entity whose two manifestations are deep vein thrombosis (DVT) and pulmonary embolism (PE). After an acute PE, almost half of the patients complain residual dyspnea, despite well-conducted curative anticoagulation. Some will present persistent defects on lung scan-scintigraphy, without pulmonary hypertension. This condition defines Chronic-Thrombo-Embolic Disease(CTED). The prevalence of CTED after PE is poorly known as are its risk factors.

The primary objective is to determine the prevalence of CTED at 3 or 6 months, depending on the provoked or unprovoked character, after a PE.

The secondary objectives are:

* To determine the potential risk factors for the occurrence of CTED.
* To look for an association between the persistence of DVT and the occurrence of CTED.
* To look for an association between the diagnosis of CTED and PE recurrence during the 12-month follow-up.
* To determine the diagnostic performance of the clinician alone compared to the lung scintigraphy (gold standard) for the diagnosis of CTED.
* To compare the impact on the quality of life (QoL) with or without CTED.
* To determine the correlation between impaired QoL and the degree of residual obstruction on lung scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* definite PE with expected life expectancy of more than 3 months - Age ≥ 18 years old.
* Patients with a first episode of symptomatic pulmonary embolism, diagnosed by CT angiography or pulmonary scintigraphy and treated in a conventional manner.
* Having received oral information about the study and having expressed a non-opposition to participate to the study
* Benefiting from a social security scheme

Exclusion Criteria:

* Patients with pulmonary hypertension.
* Patients who have already had a recurrence of pulmonary embolism or deep vein thrombosis of the lower limbs.
* Patients with a contraindication to performing a lung ventilation-perfusion scintigraphy.
* Patients at high risk of recurrence of venous thromboembolic disease (severe thrombophilia or active cancer).
* Classical contraindications to anticoagulants.
* Vulnerable patients: pregnant women, under guardianship or curatorship
* Premature termination of participation
* Recurrent pulmonary embolism diagnosed by CT angiography, or deep vein thrombosis diagnosed by venous Doppler ultrasound of the lower limbs within the first 3 or 6 months depending on the nature of the VTE.
* Occurence of pulmonary hypertension detected by trans-thoracic ultrasound (systolic pulmonary arterial pressure more than 35 mmgh).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all PE hospitalized for a pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Chronic thrombo-embolic disease (CTED) prevalence | 3 to 6 months after pulmonary embolism
  CTED is determined by lung ventilation-perfusion scintigraphy witch detect a persistant obstruction more than 10% of the pulmonary arteries perfusion (defined by amputation of at least two pulmonary segments on V/ Q lung scan).

SECONDARY OUTCOMES:
Associated risk factors for CTED occurrence | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: (age, BMI, D-dimer level, clinical severity-PESI score, diameter of the right ventricle on ultrasound (mm), quality ofsystolic function right ventricle on ultrasound, thrombolytic treatment, size of the pulmonary artery trunk, unprovoked nature of VTE, time between onset of symptoms and diagnosis) global clinical Data in the medical document
Associated risk factors for CTED occurrence BMI | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: BMI (kg / m²)
Associated risk factors for CTED occurrence D-dimer level | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: D-dimer level (ng / ml) on arrival
Associated risk factors for CTED occurrence clinical severity | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: clinical severity according to ESC criteria
Associated risk factors for CTED occurrence ultrasound parameters of RV function | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: clinical severity: ultrasound parameters of RV function
Associated risk factors for CTED occurrence diameter of the pulmonary artery trunk | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: clinical severity: diameter of the pulmonary artery trunk (mm) measured on ultrasound and / or CT scan
Associated risk factors for CTED occurrence need for thrombolytic therapy or infusion of inotropic agent | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: clinical severity: need for thrombolytic therapy or infusion of inotropic agent at the physician's discretion
Associated risk factors for CTED occurrence unprovoked nature of the event | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: clinical severity: unprovoked nature of the event at the physician's discretion
Associated risk factors for CTED occurrence time between onset of symptoms and diagnosis | 3 to 6 months after pulmonary embolism
  The initial risk factors are the classic cardiologic data: time between onset of symptoms and diagnosis (days)
Associated risk factors (deep vein thrombosis ) for CTED prevalence | 3 to 6 months after pulmonary embolism
  Number of patient with a persistence of a DVT and the persistence of deep vein thrombosis (The persistence of DVT being defined by the presence of a venous thrombus of the same location as that of the initial episode)
  Measurement of the level of CTED according to the persistence of deep vein thrombosis beyond diagnosis. The persistence of a DVT is defined by the presence at 3 or 6 months of a venous thrombus of the same location as the initial episode, among the patients who presented with a PE associated with a DVT.
Associated risk factors (new episode of PE or DVT ) for CTED occurrence | 3 to 6 months after pulmonary embolism
  Number of patients (with or without CTED) with a recurrence (new episode of PE or DVT) Recurrence of VTE is defined by defined by a new documented thromboembolic event with a non-normal d-dimers level.
Associated risk factors (clinical presumption of CTED ) for CTED occurrence | 3 to 6 months after pulmonary embolism
  Agreement between the clinical presumption of CTED by an experienced physician (questioning and evaluation of dyspnea) compared to the diagnosis of CTED by lung scintigraphy. The clinical presumption by the clinician (presence or not of an CTED) is based on the questioning, the clinical examination and the realization of an echocardiography, if necessary, in order to rule out pulmonary hypertension.
quality of life score | 3 to 6 months after pulmonary embolism
  Assessment of quality of life using the PembQOL score

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided